CLINICAL TRIAL: NCT07202026
Title: Patient Perspectives on Prescription Opioid Discontinuation: Understanding and Promoting Safe Transitions
Brief Title: Prescription Opioid Discontinuation: Honoring Patient Insights and Experience to Support Safe and Caring Transitions -- Decision Aid Pilot
Acronym: PHOENIX
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of Arkansas (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Clarissa Hsu, Associate Investigator, Kaiser Permanente
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R01HS027790 (AHRQ); R01HS027790 (AHRQ)
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Opioid Tapering
Keywords: Chronic pain; Decision Aids; Long-term opioid therapy; Opioid tapering
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision Aid Pilot Test (Experimental)
  Interventions: Behavioral: Patient-centered Decision Aid to support long-term opioid therapy tapering

INTERVENTIONS:
Behavioral: Patient-centered Decision Aid to support long-term opioid therapy tapering — Earlier aims of this study developed a patient-centered Decision Aid (DA) that uses stories of people who benefited from discontinuing and clear explanations of evidence for key choices to decrease stigma; empower patients; increase engagement and productive interaction with providers in decision making; and reduce fear, anger and anxiety about tapering. The DA will be designed to support conversations that providers often find challenging and help providers maintain patient trust and satisfaction. Participants in the pilot test will be asked to: 1) complete a pre-DA survey, 2) review the DA, 3) have a guided conversation with a trained study interventionist with a behavioral health background who is trained on how to use the DA, and 4) complete a post-DA survey.

SUMMARY:
Because of recent policies to decrease opioid use, some people using long-term opioid therapy (LTOT) are encouraged or required to stop (discontinue) taking opioids. That has led experts to be concerned that patients whose LTOT is discontinued could have untreated pain, turn to other substance use and possibly illicit opioids, or have worsened mental health symptoms leading to suicide. To guide safer policies, guidelines, and care, this study will interview patients and doctors about discontinuing LTOT and use the results to develop a patient-centered decision aid (DA) to improve patient-provider communication around discontinuation of LTOT. Once the DA is finalized, it will be pilot tested with a group of 30 patients who are currently on LTOT. The pilot will assess DA implementation feasibility; acceptability; knowledge transfer; and ability to successfully foster positive, patient-centered conversations about opioid discontinuation.

ELIGIBILITY:
EHR-based inclusion criteria:

* age 18 or older
* LTOT in the past 18 months (LTOT is ≥60 days of ≥50 MEDs day in each of 2 consecutive 90-day periods with medication treatment for OUD excluded)

Inclusion criteria confirmed by participant

* Have been taking opioids for chronic pain for at least 6 months
* Able to speak and read English

EHR-based exclusion criteria:

* cancer diagnosis in the last 5 years (excluding non-melanoma skin cancers)
* current palliative or hospice care
* cognitive disability
* psychiatric hospitalization in the last year
* surgery in the last 6 months
* current residence in an inpatient rehabilitation or skilled nursing facility

Exclusion criteria determined by study

- participated in an interview for Aim 1 of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Acceptability of DA | 1-2 weeks
  We will use Matlock et al.'s acceptability ranking scale to assess the acceptability of the DA to patients

CONTACTS AND LOCATIONS:
Overall Officials: Clarissa W Hsu, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No